CLINICAL TRIAL: NCT06974006
Title: Integrated Monitoring for Independent Living in Rural Settings
Brief Title: Life Monitoring for Rural Older Adults
Acronym: VIVIR
Status: Recruiting | Type: Observational
Sponsor: European University Miguel de Cervantes (Other)
Responsible Party: Sponsor
Other Study IDs: PI-DOC009-VIVIR
Record Dates: First submitted 2025-04-28; First posted 2025-05-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Aged 60 Years or Older
Keywords: Older adults; Frailty; Physical fitness; Prevention
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults living in rural areas: A single cohort of older adults (≥60 years old) will be used to evaluate the ability of a specific kit to assess the health status and predict adverse events
  Interventions: Other: Devices: Kardia Mobile 6L; Omron M7 BP ; Beurer PO30; Datospir Peak-10; NUTRILAB BIA 101 BIVA® PRO; JAMAR® Smart.

INTERVENTIONS:
Other: Devices: Kardia Mobile 6L; Omron M7 BP ; Beurer PO30; Datospir Peak-10; NUTRILAB BIA 101 BIVA® PRO; JAMAR® Smart. — Use of the Kardia Mobile 6L portable device to assess electrocardiogram; Omron M7 BP for blood pressure; Beurer PO30 for oxygen saturation; Datospir Peak-10 for peak flow; NUTRILAB BIA 101 BIVA® PRO for body composition; questionnaires for the nutritional status (Mini-Nutritional Assessment, Malnutrition Universal Screening Tool), JAMAR® Smart for handgrip strength; The Short Physical Performance Battery for frailty status and fall risk; the Geriatric Depression Scale to evaluate depression status; the Fried's frailty phenotype to assess the frailty status; the International Physical Activity Questionnaire for the physical activity levels; SARC-F to identify older adults at risk of sarcopenia; and the Timed-Up and Go for mobility, walking ability and fall risk.

SUMMARY:
Aging is a biological process that is accompanied by a progressive deterioration of physical and mental abilities and leads to an increased risk of disease. In 2023, Spain will reach an all-time high aging rate of 137.7% due to the low birth rate and increasing life expectancy. In Castilla y León, 47.57% of the population lives in municipalities with fewer than 20,000 inhabitants. This percentage has decreased over the last 10 years, reflecting a clear trend towards rural exodus, and this population loss requires the development of specific measures. Spanish Law 45/2007 includes as one of its objectives the promotion of quality social services and the guarantee of access to public services for older adults. However, geographical dispersion limits the effective implementation of these services. Although Castilla y León has a good network of local clinics, medical care in many municipalities is outpatient and limited to a weekly consultation. This low frequency of face-to-face care hinders the early detection of diseases, leads to a greater number of avoidable hospitalizations and contributes to older adults isolation. Faced with this reality, the VIVIR (Integrated Monitoring for Independent Living in Rural Settings) project proposes the implementation of an innovative system for the continuous monitoring of the health status of the elderly through an advanced comprehensive assessment kit. This kit will include instruments such as electrocardiogram, blood pressure measurement, manual grip strength, assessment of physical and emotional functions, spirometry, body composition and nutritional assessment.

DETAILED DESCRIPTION:
Advances in disease prevention and treatment as well as social changes have led to an increase in life expectancy of around 10-20 years in various regions of the world since the 1950s. However, population growth and aging have led to a sharp increase in the number of older people with physical disabilities, i.e. with difficulties in performing activities of daily living. Aging is defined as a biological process characterized by an increasing accumulation of cellular and molecular damage that leads to a decrease in physical and mental abilities and thus to an increased risk of disease. Currently, more than half of the population in the European Union is 65 years old or older. Furthermore, projections for 2050 indicate a decrease in the ratio of working-age people to older people, reflecting the increasing aging of the European population. In 2023, Spain will reach the historical peak of aging with 137.7% of the population. These demographic changes are also expected to increase the number of age-related diseases and conditions, including frailty. Frailty can be defined as a syndrome caused by the combined effect of multiple age-related and associated changes. Specifically, phenotypic frailty is a validated clinical presentation that marks a distinct clinical syndrome and pathophysiology. Furthermore, the 'Frailty Index' calculates the percentage of clinically identified conditions or impairments in relation to the number of measured diseases, symptoms, signs, impairments, disabilities and functional limitations, social environment, physical activity, mental health, cognitive status, self-assessed health and, in some cases, laboratory findings. A preventive assessment together with the implementation of a care and follow-up plan can have benefits for the well-being and independence of older adults, including reduced hospital admissions, falls and long-term mortality.

ELIGIBILITY:
Inclusion Criteria:

* People living in rural areas of less than 20,000 inhabitants belonging to the Diputación de Valladolid.
* People aged 60 years or older.

Exclusion Criteria:

* People with cognitive impairment and difficulty in understanding and responding to verbal commands.
* People who have been admitted to hospital for more than or equal to one week in the last month prior to inclusion in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults (≥60 years old) with or without chronic diseases living in rural areas of Valladolid
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Electrocardiogram (ECG) | Visits 1 (Month 1), 2 (Month 2), 3 (Month 3) and 4 (Month 7)
  A 6-lead ECG will be performed using the Kardia Mobile 6L portable device (AliveCor Inc., California, USA), which is FDA approved and used in clinical practice. This device connects to an application on the phone via Bluetooth to provide instantaneous readings. To perform the measurement correctly, users are asked to sit and rest for 5 minutes. Afterwards, the user should hold the device so that the thumbs touch the upper electrodes, and the device is in direct contact with the skin of the left leg at the knee or ankle.
  The device gives a diagnosis about heart beat rhythm (e.g., normal sinoauricular rhythm, arritmia, etc.)
Blood pressure | Visits 1 (Month 1), 2 (Month 2), 3 (Month 3) and 4 (Month 7)
  An Omron M7 automatic blood pressure monitor (Omron Healthcare Co., Ltd., Kyoto, Japan) will be used to measure blood pressure. According to the recommendations of the American Heart Association, the user should sit in a comfortable chair with lumbar support for at least 5 minutes before the measurement. The participant will be asked to place both feet flat on the floor without crossing the legs and place the arm with the cuff at chest level on a table with the palm facing up. Make sure that the cuff is properly adjusted, but not too tight and touching bare skin, before starting the blood pressure measurement. The person being tested should not speak during this procedure to ensure an accurate and reliable measurement. An initial measurement will be taken on each arm to determine the arm with the highest blood pressure. Three measurements will be then taken at least one minute apart.
  The unit measure is: Millimetre of mercury (mmHg)
Oxygen saturation | Visits 1 (Month 1), 2 (Month 2), 3 (Month 3) and 4 (Month 7)
  A Beurer PO30 pulse oximeter (Beurer GmbH, Mittelstand, Germany) will be used and placed on the index or middle finger previously cleaned with alcohol. Participants are asked not to apply nail polish to their fingernails.
  Measurement results will be given in percentage of oxygen saturation (%SatO2)
Spirometry | Visits 1 (Month 1), 2 (Month 2), 3 (Month 3) and 4 (Month 7)
  An expiratory flow meter (Datospir Peak-10, Sibelmed S.A.U, Barcelona, Spain) will be used to measure peak expiratory flow. The maneuver is performed in a seated position with both feet resting on the floor, the head in a neutral position and a nose clip is used. The participant will be instructed to perform a maximal inhalation followed by a rapid exhalation, with an expiratory effort of 1 to 2 seconds. The patient will be instructed not to cough during the technique and not to flex and/or extend the cervical spine. Three maneuvers will be performed, with the highest value being used for the analysis.
  Measurement will be given in liter per minute (l/min).
Bioimpedance | Visits 1 (Month 1), 2 (Month 2), 3 (Month 3) and 4 (Month 7)
  The NUTRILAB BIA 101 BIVA® PRO bioimpedance device (AKERN Srl, Florence, Italy) will be used. This non-invasive method measures the body's resistance and reactance of the body to the passage of a low-intensity electric current and enables the determination of various body parameters. Bioimpedance provides accurate data on body fat percentage, muscle mass, total body water and other relevant indicators such as phase angle and Z-score. Users will be instructed to remove all metal-containing objects and remain in a supine position on a couch during the measurements, with the legs in 45° abduction, the shoulders in 30° abduction relative to the center of the body and the hands in pronation. After cleaning the skin with alcohol, two adhesive electrodes (Biatrodes Akern Srl, Florence, Italy) will be placed on the surface of the right hand and two on the right foot.
  The measurement results will be given in different unit measures depending on the specific variable assessed.
Nutritional assessment | Visits 1 (Month 1), 2 (Month 2), 3 (Month 3) and 4 (Month 7)
  * Mini-Nutritional Assessment (MNA): is a screening tool that helps to identify malnourished older people or those at risk of malnutrition. It assesses 17 items and consists of two main sections, a screening and an overall assessment. The maximum total score is 30 points, with higher scores indicating better nutritional status.
  * Malnutrition Universal Screening Tool (MUST): a five-step screening tool that assesses three variables (body mass index (BMI), weight loss in 3-6 months and the impact of acute illness) to identify malnourished adults, adults at risk of malnutrition (undernutrition) or obese adults. This tool is recommended by ESPEN for adults in the community, although it is also suitable for nursing home residents and hospital patients and can be used by all health professionals. This screening serves as a predictor of hospital admissions, mortality and associated costs.
Handgrip strength | Visits 1 (Month 1), 2 (Month 2), 3 (Month 3) and 4 (Month 7)
  Handgrip strength will be assessed using the hand-held Jamar® Plus Smart Dynamometer (Patterson Medical Ltd., Sammons Preston, Nottinghamshire, UK). Manual grip strength will be recorded on both limbs and the dynamometer will be adjusted to hand size prior to testing. The participant's elbow should be in 90° flexion, the forearm is fully supported on a rigid surface (stretcher or table) and the shoulder is in a neutral position. Participants will be instructed to keep the flexion and extension of the wrist neutral. Three measurements will be taken with a one-minute break in between and the best one is used for the analysis.
  Measurements will be given in kilograms.
Short Physical Performance Battery (SPPB) | Visits 1, 2, 3 and 4
  is an instrument to assess the risk of frailty and the risk of falls. This test consists of three tests: a) balance tests; b) 4-meter walking speed; c) five-times stand-up and sit-down test (5STS). In the balance tests, participants will be asked to stand with their feet side by side for 10 seconds, then advance to walk in a half-tandem position for 10 seconds and finally to walk in a tandem position for 10 seconds or longer. For gait speed scoring, participants will be instructed to complete two 4-meter walks at their normal pace, with the faster of the two times being recorded for scoring. For the 5STS, participants are asked to cross their arms over their chest and stand and sit on a chair five times as fast as possible. Each item will be scored on a scale of 0 to 4 points, with a possible total possible score of 12 points, with higher scores indicating better physical performance.

SECONDARY OUTCOMES:
Frailty phenotype | Visits 1 (Month 1), 2 (Month 2), 3 (Month 3) and 4 (Month 7)
  The Fried frailty phenotype will be used to assess frailty status, which is composed of five main components: i) involuntary weight loss; ii) fatigue or exhaustion; iii) weakness; iv) walking speed; v) physical activity levels.
  Within this tool and with the intention of assessing physical activity levels, the International Physical Activity Questionnaire (IPAQ) will be used. This questionnaire consists of 7 questions about the frequency, duration and intensity of activity (moderate and intense) performed in the last seven days, as well as walking and sitting time in a working day. This tool allows a standardized and valid measurement of physical activity and is useful in both research and public health.
  Measurements will be given in a global score (0-5).
Sarcopenia detection | Visits 1 (Month 1), 2 (Month 2), 3 (Month 3) and 4 (Month 7)
  The risk of sarcopenia will be assessed using the most updated criteria of the European Working Group on Sarcopenia in the Elderly (EWGSOP 2). Following the algorithm proposed by them, the following assessments will be performed:
  * SARC-F: this five-question questionnaire will be used to identify subjects at risk of sarcopenia.
  * Manual grip strength: using the protocol previously described.
  * Five times sit-to-stand test: this is included in the SPPB.
  * Appendicular muscle mass: will be identified through bioimpedance performed through the protocol described above.
  * Gait speed.
  Measurements will be given in a total score and the specific results obtained in each assessment (kilograms for handgrip assessment, time (seconds) for five times sit-to-stand, total appendicular muscle mass; velocity (m/s) for gait speed; and time (seconds) for Timed Up and Go).

OTHER OUTCOMES:
Telephone follow-up | Phone calls every two weeks during the seven months of study
  This will be carried out every two weeks during the seven months of the study using a semi-structured interview to record the number of cardiovascular events, hospitalizations and falls of each participant.
  All measurements will be taken during the monthly evaluations scheduled for the first three months and seven months after the start of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Susana López Ortiz, PhD, Principal Investigator — Miguel de Cervanyes European University
Locations (1):
- Miguel de Cervantes European University, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Roman Vinas B, Ribas Barba L, Ngo J, Serra Majem L. [Validity of the international physical activity questionnaire in the Catalan population (Spain)]. Gac Sanit. 2013 May-Jun;27(3):254-7. doi: 10.1016/j.gaceta.2012.05.013. Epub 2012 Oct 24. Spanish. PMID 23103093
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Ortega Orcos R, Salinero Fort MA, Kazemzadeh Khajoui A, Vidal Aparicio S, de Dios del Valle R. [Validation of 5 and 15 items Spanish version of the geriatric depression scale in elderly subjects in primary health care setting]. Rev Clin Esp. 2007 Dec;207(11):559-62. doi: 10.1157/13111585. Spanish. PMID 18021644
- [Background] Kameniar K, Mackintosh S, Van Kessel G, Kumar S. The Psychometric Properties of the Short Physical Performance Battery to Assess Physical Performance in Older Adults: A Systematic Review. J Geriatr Phys Ther. 2024 Jan-Mar 01;47(1):43-54. doi: 10.1519/JPT.0000000000000337. Epub 2022 Apr 19. PMID 35442231
- [Background] Guigoz Y, Vellas B. Nutritional Assessment in Older Adults : MNA(R) 25 years of a Screening Tool and a Reference Standard for Care and Research; What Next? J Nutr Health Aging. 2021;25(4):528-583. doi: 10.1007/s12603-021-1601-y. PMID 33786572
- [Background] Campa F, Bongiovanni T, Rossi A, Cerullo G, Casolo A, Martera G, Trecroci A, Moro T, Paoli A. Athletic bioimpedance-based equations underestimate fat free mass components in male elite soccer players: development and validation of new soccer-specific predictive models. J Transl Med. 2023 Dec 15;21(1):912. doi: 10.1186/s12967-023-04795-z. PMID 38102652
- [Background] Magave JA, Bezerra SJS, Matos AP, Pinto ACPN, Pegorari MS, Ohara DG. Peak Expiratory Flow as an Index of Frailty Syndrome in Older Adults: A Cross-Sectional Study. J Nutr Health Aging. 2020;24(9):993-998. doi: 10.1007/s12603-020-1423-3. PMID 33155627
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] Koltowski L, Balsam P, Glowczynska R, Rokicki JK, Peller M, Maksym J, Blicharz L, Maciejewski K, Niedziela M, Opolski G, Grabowski M. Kardia Mobile applicability in clinical practice: A comparison of Kardia Mobile and standard 12-lead electrocardiogram records in 100 consecutive patients of a tertiary cardiovascular care center. Cardiol J. 2021;28(4):543-548. doi: 10.5603/CJ.a2019.0001. Epub 2019 Jan 15. PMID 30644079
- [Background] Fried LP, Cohen AA, Xue QL, Walston J, Bandeen-Roche K, Varadhan R. The physical frailty syndrome as a transition from homeostatic symphony to cacophony. Nat Aging. 2021 Jan;1(1):36-46. doi: 10.1038/s43587-020-00017-z. Epub 2021 Jan 14. PMID 34476409
- [Background] Camera A, Tabetah M, Castaneda V, Kim J, Galsinh AS, Haro-Vinueza A, Salinas I, Seylani A, Arif S, Das S, Mori MA, Carano A, de Oliveira LC, Muratani M, Barker R, Zaksas V, Goel C, Dimokidis E, Taylor DM, Jeong J, Overbey E, Meydan C, Porterfield DM, Diaz JE, Caicedo A, Schisler JC, Laiakis EC, Mason CE, Kim MS, Karouia F, Szewczyk NJ, Beheshti A. Aging and putative frailty biomarkers are altered by spaceflight. Sci Rep. 2024 Jun 11;14(1):13098. doi: 10.1038/s41598-024-57948-5. PMID 38862573
- [Background] The Lancet Regional Health-Europe. Securing the future of Europe's ageing population by 2050. Lancet Reg Health Eur. 2023 Dec 1;35:100807. doi: 10.1016/j.lanepe.2023.100807. eCollection 2023 Dec. No abstract available. PMID 38115962
- [Background] Lisko I, Kulmala J, Annetorp M, Ngandu T, Mangialasche F, Kivipelto M. How can dementia and disability be prevented in older adults: where are we today and where are we going? J Intern Med. 2021 Jun;289(6):807-830. doi: 10.1111/joim.13227. Epub 2021 Jan 10. PMID 33314384
- See also: World Health Organization — https://www.who.int/news-room/fact-sheets/detail/ageing-and-health